CLINICAL TRIAL: NCT01680289
Title: Influence of the Number of Layers of a One Bottle Adhesive on the Longevity of Composite Resin Restorations in Primary Molars - Randomized Controlled Clinical Study.
Brief Title: Influence of the Number of Layers of a One Bottle Adhesive on the Longevity of Composite Restorations in Primary Molars
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidade Federal do Rio de Janeiro (Other)
Responsible Party: Principal Investigator, Marlus Roberto Rodrigues Cajazeira, Assistant Professor, Universidade Federal do Rio de Janeiro
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: Adhesive1; PRIMEBOND21 (Registry Identifier: Primebond)
Record Dates: First submitted 2012-08-29; First posted 2012-09-07 (Estimated); Last update posted 2014-12-02 (Estimated); Status verified 2012-09

CONDITIONS: Dental Caries; Secondary Dental Caries
Keywords: Dentin bonding agents; Composite restorations; Dental restoration failure
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Three adhesive coats (Experimental): Consecutive application of three one-bottle adhesive coats
  Interventions: Procedure: Two adhesive coats
- Two adhesive coats (Active Comparator): Consecutive application of two one-bottle adhesive coats
  Interventions: Procedure: Three adhesive coats

INTERVENTIONS:
Procedure: Three adhesive coats — After caries removal, enamel margins will be conditioned with phosphoric acid gel 37% by 15 seconds and dentin walls by 8 seconds. The etchant will be removed with use of water spray by 30 seconds. The water excess will be removed with a cotton pellet. The first layer of Prime & Bond 2.1 adhesive will be applied with a microbrush. After 20 seconds a second layer will be applied and after a similar period a third layer will be applied over cavity walls. Again, after 20 seconds, the layers will be gently air-dried and photopolymerized by 10 seconds with a LED photoactivation unit.
  Arms: Two adhesive coats
Procedure: Two adhesive coats — After caries removal, enamel margins will be conditioned with phosphoric acid gel 37% by 15 seconds and dentin walls by 8 seconds. The etchant will be removed with use of water spray by 30 seconds. The water excess will be removed with a cotton pellet. The first layer of Prime & Bond 2.1 adhesive will be applied with a microbrush. After 20 seconds a second layer will be applied and after 20 seconds, the layers will be gently air-dried by 5 seconds. The two layers will be photopolymerized by 10 seconds with a LED photoactivation unit.
  Arms: Three adhesive coats

SUMMARY:
The aim of this study is to determinate the influence of an alternative adhesive application protocol (i.e. consecutive application of an extra adhesive layer)on restoration longevity in primary molars.

DETAILED DESCRIPTION:
Adhesive systems based on total etch technique remains the most popular products among dental practitioners. These systems are based on the use of an acid conditioner to remove the smear layer and demineralize the enamel and dentin. After the removal of the conditioner by rinsing, a mixture containing the primer and adhesive - i.e. one bottle adhesives - is applicated over the demineralized tissues. The polymerization of the adhesive monomers into microporosities created by acid conditioning forms the structure knowing as hybrid layer or resin-dentin interdifusion zone. A common problem related to total etch technique is the incomplete infiltration of adhesive monomers through demineralized dentin, resulting in the presence of a zone of unprotected collagen fibrils beneath the hybrid layer that is prone to enzymatic degradation. According to some laboratory studies, consecutive application of multiple adhesive coats results in quantitative and qualitative improvements in dental adhesion. In addition to increasing the values of bond strength to dentin, consecutive application of multiple adhesive layers enhances the infiltration of adehesive monomers through demineralized dentin, resulting in a more homogenous hybrid layer.

ELIGIBILITY:
Inclusion Criteria:

* Presence of two or more pairs of caries lesions in occlusal or occluso-approximal surfaces of primary molars

Exclusion Criteria:

* Systemic diseases in which dental treatment is a risk to patient's life
* Bruxism
* Orthodontic appliance
* Absence of occlusal contact in eligible teeth
* Signs and symptoms of pulp infflamation or necrosis

Ages: 5 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2012-08; Primary Completion 2015-08 (Estimated); Study Completion 2015-08 (Estimated)

PRIMARY OUTCOMES:
Survival rate | 06, 12, 18, 24, 30 and 36 months
  Survival rate considering failure of restorations due: partial or complete loss of restorative material; marginal ditching; superficial or marginal discoloration; secondary caries; pulpal complications; wear of restorative material; tooth fracture.

SECONDARY OUTCOMES:
Marginal adaptation | 06, 12, 18, 24, 30 and 36 months
  Evaluation of resin replicas of restored teeth on scanning electron microscopy (SEM)

CONTACTS AND LOCATIONS:
Overall Officials: Marlus RR Cajazeira, MsD, Principal Investigator — Universidade Federal do Rio de Janeiro; Lucianne Cople Maia, PhD, Study Chair — Universidade Federal do Rio de Janeiro; Eduardo M da Silva, PhD, Study Chair — Universidade Federal Fluminense; Alessandro D Loguércio, PhD, Study Chair — Universidade Estadual de Ponta Grossa; Michelle M Amari, MsD, Study Director — Universidade Federal Fluminense
Locations (1):
- School of Dentistry of Federal University of Rio de Janeiro, Rio de Janeiro, Rio de Janeiro, Brazil

REFERENCES:
- [Background] Hashimoto M, Sano H, Yoshida E, Hori M, Kaga M, Oguchi H, Pashley DH. Effects of multiple adhesive coatings on dentin bonding. Oper Dent. 2004 Jul-Aug;29(4):416-23. PMID 15279481
- [Background] Hashimoto M, De Munck J, Ito S, Sano H, Kaga M, Oguchi H, Van Meerbeek B, Pashley DH. In vitro effect of nanoleakage expression on resin-dentin bond strengths analyzed by microtensile bond test, SEM/EDX and TEM. Biomaterials. 2004 Nov;25(25):5565-74. doi: 10.1016/j.biomaterials.2004.01.009. PMID 15159072
- [Background] Hashimoto M. A review--micromorphological evidence of degradation in resin-dentin bonds and potential preventional solutions. J Biomed Mater Res B Appl Biomater. 2010 Jan;92(1):268-80. doi: 10.1002/jbm.b.31535. PMID 19904824
- [Background] Pashley DH, Tay FR, Yiu C, Hashimoto M, Breschi L, Carvalho RM, Ito S. Collagen degradation by host-derived enzymes during aging. J Dent Res. 2004 Mar;83(3):216-21. doi: 10.1177/154405910408300306. PMID 14981122
- [Background] Hashimoto M, Ohno H, Kaga M, Sano H, Endo K, Oguchi H. The extent to which resin can infiltrate dentin by acetone-based adhesives. J Dent Res. 2002 Jan;81(1):74-8. doi: 10.1177/002203450208100116. PMID 11820372
- See also: School of Dentistry of Federal University of Rio de Janeiro web site — http://www.odontologia.ufrj.br